CLINICAL TRIAL: NCT07065786
Title: A Generative Model-based System for Predicting Survival and Guiding Treatment Decisions in Patients With Unresectable Hepatocellular Carcinoma Undergoing Transarterial Chemoembolization in Combination With Immunotherapy and Targeted Therapy
Brief Title: A Generative Model-based System for Predicting Survival and Guiding Treatment Decisions in Patients With Unresectable Hepatocellularcarcinoma Undergoing Transcatheter Arterial Chemoembolization in Combination With Immunotherapy and Targeted Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Professor of Radiology Zhongda Hospital, Southeast University, Zhongda Hospital
Other Study IDs: GenTI-uHCC
Record Dates: First submitted 2025-07-01; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Transcatheter Arterial Chemoembolization; Unresectable Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; gengerative model; transcatheter arterial chemoembolization; immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- development cohort, validation cohort, test cohort
  Interventions: Other: Generative model

INTERVENTIONS:
Other: Generative model — Prospectively enroll pretreatment imaging data from patients with unresectable hepatocellular carcinoma undergoing TACE in combination with immunotherapy plus targeted therapy. Utilize a generative model to create virtual images that represent optimal treatment responses, and compare these virtual images with actual treatment response images collected during follow-up to evaluate the reliability of the generative model.

SUMMARY:
The entry point of this study is the proposition of "generative longitudinal prediction," which utilizes only pre-treatment imaging to create high-fidelity predictions of post-treatment imaging. This approach effectively overcomes the clinical challenge of acquiring genuine longitudinal follow-up data. This paradigm shift not only tackles the scarcity of longitudinal data but also introduces an innovative method for treatment simulation using digital twins. Clinicians can intuitively assess the potential efficacy of various treatment plans before intervention through virtually generated multi-timepoint imaging, providing a visual foundation for personalized treatment decisions. This research merges generative AI with dynamic risk models to achieve: 1) a transition from static assessment to dynamic simulation; 2) earlier survival predictions; and 3) personalized optimization of treatment plans. By eliminating dependence on longitudinal data, we aim to deliver more precise and individualized treatment decision support for advanced liver cancer patients, ultimately enhancing survival outcomes and quality of life.

DETAILED DESCRIPTION:
The entry point of this study is the proposition of "generative longitudinal prediction," which utilizes only pre-treatment imaging to create high-fidelity predictions of post-treatment imaging. This approach effectively overcomes the clinical challenge of acquiring genuine longitudinal follow-up data. This paradigm shift not only tackles the scarcity of longitudinal data but also introduces an innovative method for treatment simulation using digital twins. Clinicians can intuitively assess the potential efficacy of various treatment plans before intervention through virtually generated multi-timepoint imaging, providing a visual foundation for personalized treatment decisions. This research merges generative AI with dynamic risk models to achieve: 1) a transition from static assessment to dynamic simulation; 2) earlier survival predictions; and 3) personalized optimization of treatment plans. By eliminating dependence on longitudinal data, we aim to deliver more precise and individualized treatment decision support for advanced liver cancer patients, ultimately enhancing survival outcomes and quality of life. The model was developed in a retrospective cohort, with validation and testing conducted in multiple retrospective and prospective cohorts, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as unresectable hepatocellular carcinoma (HCC) by histopathology and/or clinical diagnosis (typical imaging features, clinical manifestations, laboratory tests, etc.) (Reference: Guidelines for Diagnosis and Treatment of Primary Liver Cancer (2024 Edition));
* Patients with unresectable HCC receiving TACE combined with targeted immunotherapy;
* Liver function classified as Child-Pugh A or B;
* Aged 18 or above, regardless of gender;
* Expected survival time ≥3 months;
* ECOG PS score ≤2;
* Meeting the following laboratory parameters: a) Hematologic function: Absolute neutrophil count ≥1.0×10⁹/L; Platelet count ≥50×10⁹/L; Hemoglobin ≥90 g/L; International normalized ratio (INR) <1.7 or prothrombin time prolongation ≤4 seconds; b) Liver function: ALT/AST ≤5× upper limit of normal (ULN); Total bilirubin ≤210 μmol/L [≤2.38 mg/dL]; Albumin ≥28 g/L; c) Renal function: Serum creatinine ≤1.5× ULN.

Exclusion Criteria:

* Concurrent presence of other malignant tumors besides HCC;
* Moderate to severe ascites (ascites scoring 3 points on the Child-Pugh scale); - - Receipt of other first-line, second-line, or third-line systemic therapies (including any regimen of systemic treatment) or any local therapies (including transcatheter interventional therapy, ablation therapy, internal/external radiotherapy, etc.), as well as surgical resection or herbal medicine within 4 weeks prior to TACE combined with targeted immunotherapy;
* Incomplete data, such as missing baseline laboratory test results, unavailable or poor-quality imaging data, or lack of prognostic information;
* Severe liver dysfunction: e.g., decompensated cirrhosis or other liver diseases significantly affecting bilirubin levels;
* Severe comorbidities: e.g., refractory hypertension (blood pressure remaining above 150/100 mm Hg despite optimal medication), persistent arrhythmia (CTCAE grade 2 or higher), atrial fibrillation of any degree, prolonged QTc interval (>450 ms in males or >470 ms in females), renal insufficiency, etc.;
* Co-infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS);
* Pregnant or breastfeeding women;
* Acute or chronic psychiatric disorders (including those affecting participant enrollment, treatment intervention, or follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable hepatocellular carcinoma undergoing TACE in combination with immunotherapy plus targeted therapy
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Through study completion, an average of 20 months
  defined as the time from the initial of combined therapy to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT07065786/Prot_000.pdf